CLINICAL TRIAL: NCT07401875
Title: A Phase 1b Study of HC-7366, an Agonist of ISR With Immunotherapy in Kidney Cancer (SHARK)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1590; NCI-2026-00890 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Phase 1b; HC-7366; SHARK; Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doublet Cohort (Experimental): Treatment with Nivolumab + HC-7366 (PO) Q4W
  Interventions: Drug: Nivolumab; Drug: HC-7366
- Triplet Cohort (Experimental): Treatment with Nivolumab + Ipilimumab + HC-7366 (PO) Q4W
  Interventions: Drug: Nivolumab; Drug: HC-7366; Drug: ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Given by IV
Drug: HC-7366 — Given by po
Drug: ipilimumab — Given by IV
  Arms: Triplet Cohort

SUMMARY:
To find out if the combination of HC-7366 and nivolumab (with or without ipilimumab) can help to control ccRCC. The

DETAILED DESCRIPTION:
Primary Objectives

To assess two combinations of HC-7366:

* Doublet Cohort: HC-7366 with nivolumab monotherapy
* Triplet Cohort: HC-7366 with nivolumab/ipilimumab dual immune checkpoint inhibition

  * For safety through assessment of trial-limiting toxicities including need for high dose corticosteroids (= 40 mg prednisone equivalents for two weeks or more)
  * For antitumor activity through assessment of Overall response rate (ORR) and Disease control rate (DCR: CR or partial response (PR) or stable disease (SD)) per RECIST v1.1

Secondary Objectives The secondary objectives of the study are to estimate median progression free survival (mPFS) and PFS at six months, duration of response (DOR), primary PD rate (progressive disease as best response), Time to response (TTR), overall survival (OS) median and at one year, immune related Adverse Event (irAE) rate, and to evaluate participant reported outcomes using the FKSI-23 and the FACT-ICM Subscale.

ELIGIBILITY:
Eligibility Criteria

1. Ability to understand and the willingness to sign a written informed consent document
2. Male or female ≥ 18 years of age
3. Confirmed diagnosis of clear cell RCC
4. Stage IV metastatic RCC per American Joint Committee on Cancer
5. Triplet Cohort (IO/IO): No prior systemic therapy for advanced RCC or prior adjuvant therapy allowed.
6. Doublet Cohort: Participant must have progressed on at least one PD1 based doublet regimen (IO/IO or IO/TKI). Prior adjuvant therapy is allowed and does count as one line of systemic therapy.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 )
8. At least one measurable lesion as defined by RECIST 1.1

   • A tumor lesion situated in a previously irradiated area is considered a measurable/target lesion only if subsequent disease progression has been documented in the lesion
9. Has pathology-confirmed RCC. Extra tissue should be submitted if available for correlatives. Formalin-fixed paraffin-embedded tissue blocks are preferred to slides. Details pertaining to tumor tissue submission can be found in the Lab Procedures Manual.
10. Willing and able to undergo bone and brain scans at baseline and continue to have scans performed if positive at screening.
11. Adequate organ function within 28 days prior to first dose of protocol-indicated treatment, including:

    * White blood cell (WBC) ≥ 2,000 /μL
    * Absolute neutrophil count (ANC) ≥ 1,000/μL
    * Platelet count ≥ 100,000/μL
    * Hemoglobin (Hgb) ≥ 9.0 g/dL in prior 4 weeks. Blood transfusions are allowed to achieve this.
    * Serum creatinine ≤ upper limit of normal (ULN), or calculated creatinine clearance ≥ 30 mL/min (per the Cockcroft-Gault formula,)
    * Total bilirubin ≤ ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 3.0 mg/dL)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN
12. Women must not be breastfeeding while taking the study drug and for up to five months after the last dose of study drug
13. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to receiving first dose of protocol-indicated treatment

    * "Women of childbearing potential" (WOCBP) is defined as any female who has experienced menarche who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal
    * Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological causes
    * If menopausal status is considered for the purpose of evaluating childbearing potential, women < 62 years of age must have a documented serum follicle stimulating hormone (FSH) level within laboratory reference range for postmenopausal women, in order to be considered postmenopausal and not of childbearing potential
14. Women of childbearing potential (WOCBP) must agree to follow instructions for acceptable contraception prior to the study and from the time of signing consent, for the duration of the study participation and for 23 weeks after their last dose of protocol-indicated treatment

    * The effects of HC-7366 on the developing human fetus are unknown. For this reason and because first-in-class, first-in-human agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114).
    * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the study and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
15. Men not azoospermic who are sexually active with WOCBP must agree to follow instructions for acceptable contraception prior to the study and from the time of signing consent, for the duration of the study participation, and for 31 weeks after their last dose of protocol-indicated treatment
16. Participant s with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
17. Participant s with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
18. Participant s with previously treated brain metastases may be eligible provided they are radiologically (by MRI) and clinically stable (i.e., without evidence of disease progression) for at least 4 weeks (28 days) by repeat imaging (repeat imaging should be performed during study screening), with no evidence of new or enlarging brain metastases, and without requirement for steroid treatment for at least 28 days prior to the first dose of study drug or study therapy. (CT is acceptable if MRI is contraindicated)
19. Participant s with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this study
20. Participant s with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this study, participant s should be class 2B or better

Exclusion Criteria

1. For the Triplet Cohort (Nivo/Ipi/HC-7366):

* Prior systemic treatment including neoadjuvant or adjuvant therapy including an immune checkpoint inhibitor or TKI 2. For the Doublet Cohort (Nivo/HC-7366):
* More than 3 prior lines of systemic therapy allowed
* Has received any type of small molecule kinase inhibitor (including investigational kinase inhibitor) ≤ 2 weeks before start of study drug or study therapy 3. ≤ 28 days before first dose of protocol-indicated treatment:
* Major surgery requiring general anesthesia 4. ≤ 14 days before first dose of protocol-indicated treatment:
* Radiosurgery or radiotherapy
* Minor surgery. (Note: Placement of a vascular access device is not considered minor or major surgery)
* Active infection requiring systemic treatment 5. Known or suspected clinically significant active bleeding including active hemoptysis 6. Inability to swallow oral medication; or the presence of a poorly controlled gastrointestinal disorder that could significantly affect the absorption of oral study drug - e.g. Crohn's disease, ulcerative colitis, chronic diarrhea (defined as > 4 loose stools per day), malabsorption, or bowel obstruction 7. Central nervous system (CNS) metastasis, unless asymptomatic and radiologically (by MRI) and clinically stable (i.e., without evidence of disease progression) for at least 4 weeks (28 days) by repeat imaging (repeat imaging should be performed during study screening), with no evidence of new or enlarging brain metastases, and without requirement for steroid treatment for at least 28 days prior to the first dose of study drug or study therapy. (CT is acceptable if MRI is contraindicated 8. Any condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone or equivalent daily) or other immunosuppressive medications within 14 days prior to initiating protocol-indicated treatment
* In the absence of active autoimmune disease: Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intraarticular, intranasal, and inhalational) ≤ 10 mg/day prednisone or equivalent daily; and physiologic replacement doses of systemic corticosteroids ≤ 10 mg/day prednisone or equivalent daily (e.g. hormone replacement therapy needed in participants with hypophysitis) 9. Active, known or suspected autoimmune disease
* Subjects with type I diabetes mellitus; hypothyroidism only requiring hormone replacement; skin disorders such as vitiligo, psoriasis or alopecia not requiring systemic treatment; or conditions not expected by the investigator to recur in the absence of an external trigger are permitted to enroll 10. Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the investigator to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with and interpretation of scheduled visits, treatment schedule, laboratory tests and other study requirements 11. Pregnant women are excluded from this study because HC-7366 is novel, first-in-class small molecule agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with HC-7366, breastfeeding should be discontinued if the mother is treated with HC-7366. These potential risks may also apply to other agents used in this study 12. Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this study 13. Participants who are receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-07-28 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org